CLINICAL TRIAL: NCT03175991
Title: Gynacological Imaging Reporting and Data System in Classifying Ovarian Masses on the Basis of Ultrasonography
Brief Title: Gynacological Imaging Reporting and Data System in Ovarian Masses by Ultrasonography
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hagar Desoky, Principle investigator, Assiut University
Other Study IDs: HAGAR098765
Record Dates: First submitted 2017-05-29; First posted 2017-06-05 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ovarian masses patients: women of different age groups diagnosed as having an ovarian mass or accidentally discovered ovarian mass in non-complaining female by ultrasonography or Patients known to have primary that may give metastasis to the ovaries.
  Interventions: Diagnostic Test: ultrasonography

INTERVENTIONS:
Diagnostic Test: ultrasonography — A morphologic evaluation will be performed according to International Ovarian Tumor Analysis Group recommendations for the following parameters:
  Bilaterality , wall thickness, septations , papillary projections, solid areas, and echogenicity. The presence of ascites also will be recorded. Pattern recognition analysis will be used for ovarian masses highly suggestive of some diseases , then color Doppler will be activated to identify vascular color signals within the lesion.

SUMMARY:
Ovarian masses are common problems in clinical practice. Sonography is considered the firstline imaging technique for discriminating between malignant and benign lesions, and it has been shown to be useful for determining optimal treatment.

DETAILED DESCRIPTION:
Transvaginal Ultrasonography has been demonstrated to be the most sensitive and effective technique, being also non-invasive and in-expensive maneuver.Since in early reports, a standardized method for the description of the sonographic appearance of the ovarian masses was not used, the data of different studies are not easily compared.

In addition, there is no consensus on sonographic diagnostic criteria for ovarian cancer, despite many ultrasonography features being considered to be predictive of malignancy, such as presence of septations, internal nodularity, wall thickening, solid areas, free fluid or bilaterality.Usually the clinical management decision is based on data provided in the sonographic report. Many sonographers and sonologists use scoring systems to characterize ovarian masses, whereas others use the so called pattern recognition approach However, sometimes sonographic reports are misleading and confusing for the clinician. Although some groups have made considerable efforts in establishing terms and definitions for sonographic findings in ovarian masses .

In this study, we proposed a new data reporting system for sonographic findings in ovarian masses. This system is based on the concept developed for breast imaging, namely the Breast Imaging Reporting and Data System classification. Originally developed for mammographic findings, it has been successfully applied to breast sonography.

Like its breast sonographic counterpart, the gynacological imaging reporting and data system in ovarian masses by ultrasonography lexicon is intended to provide a unified language for sonographic reporting and for avoiding confusion in communication between the sonographer / sonologist and the clinician..

This system is based on a description of the ovarian mass using the pattern recognition approach and color Doppler blood flow location and the prior risk for malignancy in each group. On this basis, the proposed classification enables the sonologist or sonographer to give the clinician as much information as possible in a summarized way, as well as an estimated risk of malignancy, based only on the sonographic characteristics of the images.

Currently, there is enough evidence to indicate that when an experienced examiner performs the sonographic examination, such accuracy is achievable for most types of ovarian masses.

ELIGIBILITY:
Inclusion Criteria:

* All women of different age groups diagnosed as having an ovarian mass.
* Accidentally discovered ovarian mass in non-complaining female.
* Patients known to have primary that may give metastasis to the ovaries.

Exclusion Criteria:

* Patients receive neo adjuvant chemotherapy
* Recurrent ovarian masses

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: The study will included 123 females Who referred to radiodiagnosis department at South Egypt Cancer Institute of different ages ,diagnosed as having ovarain mass
Sampling Method: Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
The resistivity index | 10 minutes
  The resistive index will be automatically calculated from at least 3 consecutive flow velocity waveforms

CONTACTS AND LOCATIONS:
Overall Officials: Lamiaa M Refaat, Lecturer, Study Director — south egypt cancer institue,assuit univeristy; hagar HM Desoky, demonstrator, Principal Investigator — south egypt cancer institue,assuit univeristy
Locations (1):
- Faculty of Medicine-Assuit Univeristy, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang T, Li F, Liu J, Zhang S. Diagnostic performance of the Gynecology Imaging Reporting and Data System for malignant adnexal masses. Int J Gynaecol Obstet. 2017 Jun;137(3):325-331. doi: 10.1002/ijgo.12153. Epub 2017 Apr 12. PMID 28295272